CLINICAL TRIAL: NCT06015646
Title: Lifestyle Education and Personalized Coaching for Fatigue Mitigation in Emergency Medicine Residents: A Pilot Study
Brief Title: Lifestyle Coaching for Fatigue Mitigation in Emergency Medicine Residents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maryam S Makowski, PhD, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-67719; 254764 (Other: The Stanford Medicine Teaching and Mentoring Academy)
Record Dates: First submitted 2023-08-05; First posted 2023-08-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lifestyle, Healthy; Sleepiness; Alertness; Shift-Work Related Sleep Disturbance; Work Related Stress; Self Efficacy; Self-Compassion
Keywords: physician well-being; occupational well-being; resident well-being; physician coaching; lifestyle coaching; night shifts
MeSH Terms: conditions — Sleepiness; Occupational Stress

STUDY DESIGN:
Intervention Model Description: The investigators will randomize the participants who have consented to participate in the study to intervention or control arms at the beginning of each of the 3-week study periods. Participants will wear a Fitbit watch for one week prior and one week after 3-4 night shifts. The baseline online survey will collect data on sex, training year, current satisfaction levels with lifestyle strategies, morning-evening chronotype, Sleep-related Impairment, and Task Load. During the nightshifts, the following outcome measures: psychomotor vigilance test, Stanford Sleepiness Scale, Task Load Index, and Noordsy-Dahle Subjective Experience Scale will be assessed during the window of circadian low (2 to 6 am) and at a time that is most convenient time for each participant. A final online survey will assess satisfaction levels with lifestyle strategies, Sleep-related Impairment, Task Load, and satisfaction and feedback about the program at the end of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: One of the two principal investigators and researchers who analyze the data will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Coaching and Educational Handout (Experimental): Lifestyle coach-led 30-minute focused, personalized session in addition to educational handout containing lifestyle tips for fatigue mitigation in night shift workers, which will be given to all participants at the beginning of the study.
  Interventions: Behavioral: Personalized lifestyle coaching and educational handout; Behavioral: Handout
- Educational Handout Control (Active Comparator): An educational handout containing lifestyle tips for fatigue mitigation in night shift workers will be given to all participants at the beginning of the study. Personalized coaching will not be offered to participants in this arm.
  Interventions: Behavioral: Handout

INTERVENTIONS:
Behavioral: Personalized lifestyle coaching and educational handout — Participants will receive a one-page educational handout on strategies to minimize fatigue at the beginning of the study. Participants will also receive a 30-minute focused, personalized lifestyle coaching within a week of the initial overnight shift. The lifestyle coach will be in close contact during the night shifts.
  Arms: Lifestyle Coaching and Educational Handout
Behavioral: Handout — Participants will receive a one-page educational handout on strategies to minimize fatigue at the beginning of the study

SUMMARY:
The purpose of this study is to determine whether personalized lifestyle coaching minimizes the negative impact of circadian disruption on performance and recovery in emergency medicine physician trainees during night shifts.

DETAILED DESCRIPTION:
The goal of this study is to examine whether a brief personalized fatigue-mitigation lifestyle coaching (PFMLC) for emergency medicine residents on overnight shifts would minimize the negative effects of circadian rhythm disruptions on performance and recovery compared to those who receive one-time passive information on lifestyle practices.

ELIGIBILITY:
Inclusion Criteria:

* Stanford Health Care (SHC) Emergency Medicine residents (PGY 1 to 4)
* Scheduled to work at least 3 consecutive overnight shifts at SHC Emergency Department.

Exclusion Criteria:

* Non-Stanford Health Care (SHC) Emergency Medicine residents
* Stanford Health Care (SHC) Emergency Medicine residents who are not rotating in Stanford Emergency Medicine Department

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean of the 3 overnight reaction time reciprocal of the psychomotor vigilance test | 3 night shifts
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by the PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  Investigators will compare the mean of the 3 overnight Mean reaction time reciprocal (lower is desirable) of the PVT tests between the control and intervention groups.
Mean of the 3 overnight number of lapses in psychomotor vigilance test | 3 night shifts
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by the PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  Investigators will compare the mean of the 3 overnight number of lapses ( lower is desirable) of the PVT test between the control and intervention groups.
Mean of the 3 overnight number of false starts in the psychomotor vigilance test | 3 night shifts
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by the PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  Investigators will compare the mean of the 3 overnight number of false starts (lower is desirable) in the PVT test between the control and intervention groups.
Mean of the 3 overnight Aggregate Scores of the psychomotor vigilance test | 3 night shifts
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by the PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  Investigators will compare the mean of the 3 overnight Aggregate Score (0 worst-100 best and derived from the number of lapses and false starts) of the PVT test between the control and intervention groups.
Mean of the 3 overnight Stanford Sleepiness Scale | 3 night shifts
  The Sleepiness Symptom Scale (SSS) is a validated subjective measure of sleepiness frequently used for research and clinical purposes. It evaluates sleepiness at specific moments in time using a single-item scale. Respondents select one of seven statements to indicate their level of perceived sleepiness. Score Range: The scale score ranges from 1 to 7, reflecting the varying degrees of sleepiness experienced by respondents. This test takes approximately 15 seconds to complete.
  Directionality: Higher scores on the SSS represent higher perceived sleepiness, while lower scores indicate increased alertness and desirable.
  Investigators will compare the mean of the 3 overnight SSS scores between the control and intervention groups
Mean of the 3 overnight Noordsy-Dahle Subjective Experience Scale (NDSE) | 3 night shifts
  Modified version of Noordsy-Dahle Subjective Experience Scale (NDSE) for healthy adults includes 8 sub-domains:
  Global well-being, Delighted 1 to Terrible 7, Lower score better Anxiety: None 1 to Extreme 7, Lower score better Depression: None 1 to Extreme 7, Lower score better Energy: Tired 1 to Energized 7, Higher score better Motivation: None 1 to Strong 7, Higher score better Clarity of thought: Clouded 1 to Totally Clear 7, Higher score better Concentration: Poor 1 to Excellent 7, Higher score better Social interest: Alone 1 to With Others 7, Higher score better
  This test takes approximately 90 seconds to complete. Investigators will compare the mean of the 3 overnight Noordsy-Dahle Subjective Experience Scale scores between the control and intervention groups.

SECONDARY OUTCOMES:
Mean of total sleep hours | 3 weeks
  Investigators will compare total sleep hours per 24-hour period during a baseline week, a night float week, and a recovery week using FitBit Versa 4, between the two groups.
Mean of heartrate variability | 3 weeks
  Investigators will compare the heart rate variability per 24-hour period during a baseline week, a night float week, and a recovery week using Fitbit Versa 4, between the two groups.

OTHER OUTCOMES:
Percentage change from baseline in NIH PROMIS Short Form Sleep-Related Impairment | 3 weeks
  The NIH PROMIS Short Form Sleep-Related Impairment Scale is included as an exploratory outcome measure in this study. The Sleep-Related Impairment is designed to assess the impact of sleep-related impairment on various aspects of daily functioning and overall quality of life. Higher scores indicate greater sleep-related impairment. It takes about 1 minute to complete and will be measured at the beginning of the study and at the end of the study. Investigators will compare the percentage change from baseline between the two groups. The minimum score is 8 and the maximum is 40 and linked to T-scores ranging from 30 to 80.1. With lower scores being more favorable.
Percentage change from baseline in Task Load Index | 3 weeks
  The National Aeronautics and Space Administration (NASA) Task Load Index (TLX) is included as an exploratory outcome measure in this study. The TLX is a measure of perceived workload and is used to measure cognitive load. Lower scores are more desirable. It takes about 1 minute to complete and will be measured at the beginning of the study and at the end of the study. Investigators will compare the percentage change from baseline between the two groups. The score ranges from 0 to 600 with lower scores being more favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Al'ai Alvarez, MD, Principal Investigator — Stanford University; Maryam S Makowski, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No